CLINICAL TRIAL: NCT00777127
Title: Long-term Effects of Aldara® 5% Cream and Solaraze® 3% Gel in the Treatment of Actinic Keratoses on the Face or Scalp (LEIDA)
Brief Title: Long-term Effects of Imiquimod and Diclofenac in Actinic Keratoses
Acronym: LEIDA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X-03016-3271; 2007-004884-24 (EudraCT Number)
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2013-01

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; invasive SCC; in situ SCC; histological classification; histological progression; clinical clearance; cryotherapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aldara 5% Cream
  Interventions: Drug: Imiquimod
- 2 (Active Comparator): Solaraze 3% Gel
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Imiquimod — One course of treatment (COT) consisting of an overnight application of IMIQ (1 sachet for up to 50 cm2), applied 3 nights per week (e.g. Monday, Wednesday, Friday) for 4 weeks followed by a 4 weeks treatment pause. If necessary, this may be followed by a second COT.
  Arms: 1
Drug: Diclofenac — Solaraze® is applied locally to the skin 2 times daily and smoothed into the skin gently. The amount needed depends on the size of the lesion. Normally 0.5 grams (the size of a pea) of the gel is used on a 25 cm2 lesion site. The duration of therapy is 12 weeks.
  Arms: 2

SUMMARY:
This clinical trial serves the purpose to compare the long-term effects of a treatment of actinic keratosis - your skin disorder - using Aldara® 5% cream or Solaraze® 3% gel on the face or the scalp. In particular, it should be found out whether the healing effect of these two medications on the skin lesions (i.e. the damaged skin parts) can be maintained for a prolonged period.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompetent patient.
* A study treatment area must be identifiable: Minimum of 5 and maximum of 10 typical visible AKs in one contiguous area of up to 50 cm2 on the face or scalp. The eyelids, the inside of the nostrils or ears, or the lip area inside the vermilion border must not be part of this area.
* A positive histological finding for AK grade I or II (see Section 7.1.1.2). This will be determined from the most suspicious lesion in the STA and there from the most pathological area biopsied during screening visit. This analysis will be done by the central histopathological laboratory.
* Willingness to comply with the obligations of the study.

Exclusion Criteria:

Safety concerns:

* History of allergic reaction to imiquimod, diclofenac, acetyl salicylic acid, other non steroidal anti-inflammatory drugs (NSAID), hyaluronic acid, or relevant excipients.
* Pregnancy, breast-feeding or planned pregnancy during the study. Women of child bearing potential not using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, tubal ligation or vasectomised partner.

Lack of suitability for the study:

* Presence of AK lesions in the STA with clinically marked hyperkeratosis or hypertrophy as seen in cutaneous horns.
* Any topical AK treatment including imiquimod or diclofenac, or any systemic AK treatment such as systemic retinoids, or any surgical AK treatment at the STA within the last 2 months prior to randomisation.
* Persisting AK lesion at screening visit following topical treatment with imiquimod or diclofenac in the STA.
* Topical treatment with imiquimod or diclofenac anywhere else on the body within the last 2 months prior to randomisation.
* Presence of any histologically confirmed skin tumour in the STA: in situ SCC including Bowen's disease, invasive SCC, basal cell carcinoma, or other malignant tumours.
* Any dermatological disease or condition that may exacerbate by treatment with imiquimod or diclofenac (e.g. rosacea, psoriasis, atopic dermatitis).
* Any dermatological disease or condition in the STA that causes difficulty with examination (e.g. eczema).
* Systemic immunomodulatory treatment such as interferon, azathioprine, cyclosporine, retinoids, any oral or injectable corticosteroids, or inhaled or nasal corticosteroids with dosages of >1200 µg/day beclomethasone or equivalent within 4 weeks before start of study treatment.
* History of any malignant tumour with high tumour burden or any systemic antitumour treatment (incl. radiotherapy).
* History of any malignant skin tumour having metastasised or where metastasis could be expected.
* History of severe cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, mental, neurological, or other disease within the last two years.
* Mentally incapacitated patient.
* Present or history of drug or alcohol abuse within the last 3 years.

Administrative reasons:

* Exposure to an investigational product within the last 3 months.
* Lack of ability or willingness to give informed consent.
* Age below 18 years.
* Lack of willingness to have personal study related data collected, archived or transmitted according to protocol.
* Anticipated non-availability for study visits/procedures.
* Vulnerable subjects (such as persons kept in detention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Recurrence with respect to the study treatment area until month 12 | week 20 until month 12
  A patient is classified as recurrent when cleared at Visit Week 20 and having later on at least one clinically diagnosed AK lesion in the study treatment area

SECONDARY OUTCOMES:
Time to recurrence | 3 years
Long-term outcome with respect to development of SCC (in situ and/or invasive) | 3 years
Need of rescue treatment | 3 years
Haematological changes | 20 weeks
Cosmetic outcome. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Harald Gollnick, MD, Prof., Principal Investigator — Otto-von-Guericke-University of Magdeburg/Germany, Clinic for Dermatology and Venereology; Ursula Petzold, PhD, Study Director — MEDA Pharma GmbH & Co. KG, Bad Homburg/Germany
Locations (26):
- Austria (4):
  - Hospital Feldkirch, Department for Dermatology and Venereology, Feldkirch
  - Medical University Graz, University Clinic for Dermatology and Venereology, Graz
  - Medical University Innsbruck, University Clinic for Dermatology and Venereology, Innsbruck
  - Medical University Vienna, Department for General Dermatology, Vienna
- France (5):
  - CHU St Jacques, Department for Dermatology, Besançon
  - Hospital Sainte Marguerite, Department for Dermatology and Venereology, Pavilion 3, First Floor, Marseille
  - CHU Nice - Hospital Archet 2, Department for Dermatology, Nice
  - Hospital Saint-Louis, Derpartment for Dermatology, Paris
  - Hospital Center Lyon South, Department for Dermatology and Immuno-Allergology, Pierre-Bénite
- Germany (17):
  - Licca Clinical Research Institute, Augsburg
  - Charite - Medicine University Berlin, Dermatoma Center, Clinic for Dermatology, Allergology and Venereology, Berlin
  - Medical Practice Dominicus / Bockhorst, Dülmen
  - Medical practice, Düsseldorf
  - University Clinic Düsseldorf, Clinic for Dermatology, Düsseldorf
  - Clinic and Medical Faculty of Johann Wolfgang Goethe-University, Center for Dermatology and Venereology, Frankfurt am Main
  - SCiderm GmbH, Hamburg
  - Medical Practice, Hanover
  - University Clinic Schleswig-Holstein, Campus Kiel, Clinic for Dermatology, Venereology and Allergology, Kiel
  - Medical Department of Otto-von-Guericke-University Magdeburg, University Clinic for Dermatology and Venereology, Magdeburg
  - Department of Dermatology J. Gutenberg-University Mainz, Clinical Research Center, Mainz
  - Science, Onco & Beauty GbR, Practice for Dermatology and Medical Cosmetics, Mönchengladbach
  - University Clinic Münster, Clinic and Polyclinic for Skin Diseases, Münster
  - Clinic University Regensburg, Clinic and Polyclinic for Dermatology, Regensburg
  - Derma Center Vechta, Vechta
  - Centrovital, Witten
  - Medical practice for Dermatology and Venerology, Wuppertal